CLINICAL TRIAL: NCT03126708
Title: A Phase II, Multicenter, Open-Label, Randomized, Controlled Study to Assess Efficacy and Safety of Cetuximab in Combination With Paclitaxel Plus Cisplatin Versus Paclitaxel Plus Cisplatin Alone for the First-line Treatment of Chinese Subjects With Metastatic Esophageal Squamous Cell Carcinoma.
Brief Title: Cetuximab in Combination With Paclitaxel Plus Cisplatin Versus Paclitaxel Plus Cisplatin Alone for the First-line Treatment of Metastatic Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Director,Department of GI Oncology,Peking University, School of Oncology, Beijing Cancer Hospital & Institute, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESCC-Cetuximab-PKU
Record Dates: First submitted 2017-04-12; First posted 2017-04-24 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Esophageal Cancer, Squamous Cell; Cetuximab Effect; Chemotherapy Effect
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Cetuximab; Cisplatin; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- chemotherapy (cisplatin plus paclitaxel) and cetuximab (Experimental)
  Interventions: Drug: cetuximab; Drug: cisplatin plus paclitaxel
- chemotherapy (cisplatin plus paclitaxel) (Active Comparator)
  Interventions: Drug: cisplatin plus paclitaxel

INTERVENTIONS:
Drug: cetuximab — cetuximab (EGFR monoclonal antibody) plus standard chemotherapy
  Arms: chemotherapy (cisplatin plus paclitaxel) and cetuximab
Drug: cisplatin plus paclitaxel — Chemotherapy

SUMMARY:
This is an open-label, randomized, controlled trial. At the end of a 28-day screening period, all eligible subjects will be randomly assigned into treatment Arm A or B in a 1:1 ratio. Subjects in Arm A will receive a maximum of 6 cycles of chemotherapy (cisplatin plus paclitaxel) and cetuximab weekly in the absence of progressive disease (PD), as assessed by the Investigator, and unacceptable toxicity. After 6 cycles of treatment, subjects who derive clinical benefit will continue treatment with cetuximab as monotherapy until either PD or unacceptable toxicity. Subjects in Arm B will receive the same chemotherapy regimen as Arm A alone for a maximum of 6 cycles in the absence of PD and unacceptable toxicity.

ELIGIBILITY:
* Inclusion Criteria:

  * Signed written informed consent.
  * Older than 18 years of age.
  * Histologically proven squamous cell carcinoma of the esophagus.
  * Metastatic ESCC, not suitable for local-regional treatment.
  * Presence of at least 1 measurable lesion according to RECIST version 1.1.
  * ECOG performance status of 0 or 1.
  * Adequate bone marrow, haptic, renal, metabolic function.
* Exclusion Criteria:

  * Prior chemotherapy in the metastasis setting.
  * Prior chemotherapy within 6 months before entering this study.
  * Previous exposure to EGFR-targeted therapy.
  * Known central nervous system metastasis and/or leptomeningeal disease.
  * Subjects with any concurrent medical condition or disease that will potentially compromise the conduct of the trial at the discretion of investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-04-10 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months

SECONDARY OUTCOMES:
Overall Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
overall response rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
Disease control rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Peking Universtiy Cancer Hospital
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China